CLINICAL TRIAL: NCT04851288
Title: Mitochondrial-targeted Antioxidant Supplementation for Improving Age-related Vascular Dysfunction in Humans
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Douglas Seals, PI, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20-0502; R01AG066730 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Aging
MeSH Terms: interventions — mitoquinone; mitoquinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MitoQ, 20 mg/day (Experimental): Each MitoQ capsule contains 20 mg of mitoquinol mesylate. Dosage: 20 mg orally per day for 3 months.
  Interventions: Dietary Supplement: MitoQ
- Placebo (Placebo Comparator): Matched placebo capsules.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MitoQ — MitoQ is a biochemically modified form of ubiquinol
  Other Names: Mitoquinol
  Arms: MitoQ, 20 mg/day
Dietary Supplement: Placebo — Each placebo capsule contains inert excipient and is identical in appearance
  Arms: Placebo

SUMMARY:
The majority of cardiovascular diseases (CVD) occur in men and women ≥60 years of age. Vascular dysfunction, including endothelial dysfunction, as assessed by reduced endothelium-dependent dilation (EDD), and stiffening of the large elastic arteries (i.e., aortic and carotid artery stiffening), is a major mechanism of increased risk of CVD in older adults. Excess production of ROS (reactive oxygen species) by mitochondria (mtROS) has emerged as a central feature of vascular oxidative stress with aging and driver of age-related vascular dysfunction. As such, identifying novel strategies to decrease mtROS and improve vascular function, to ultimately reduce the risk of age-related CVD, is an important biomedical objective.

MitoQ is a mitochondria-targeted antioxidant that accumulates at the inner mitochondrial membrane where it is optimally positioned to reduce mtROS. Preclinical findings showed that 4 weeks of oral MitoQ supplementation completely restored EDD in old mice, ameliorated mtROS-associated suppression of EDD, and was associated with reduced arterial mtROS, oxidative stress, and improved mitochondrial health. MitoQ therapy also reduced aortic stiffness in old mice. A recent small pilot study of older adults (n=20) found that supplementation with MitoQ was well-tolerated, improved endothelial function, and reduced plasma levels of oxidized low-density lipoprotein, a circulating biomarker of oxidative stress. Consistent with the preclinical findings, preliminary mechanistic assessments in subsets of subjects from the pilot study suggested that improved endothelial function with MitoQ was mediated by reduced endothelial cell mtROS production, associated reductions in tonic mtROS-related suppression of EDD, and improved mitochondrial health, linked in part to changes in circulating factors in the serum induced by chronic MitoQ supplementation. Lastly, MitoQ reduced aortic stiffness in older adults who exhibited age-related aortic stiffening at baseline.

The investigators are conducting a randomized, placebo-controlled, double-blind clinical trial to establish oral MitoQ (20 mg/day; MitoQ, Ltd.) for 3 months vs. placebo (n=56/group) for improving endothelial function in older men and women (≥60 years), and determine the mechanisms by which MitoQ improves endothelial function. The investigators will also assess the effect of MitoQ on aortic stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and over
* Ability to provide informed consent
* Willing to accept random assignment to condition
* Body mass index <40 kg/m2
* Weight stable in the prior 3 months (<2 kg weight change) and willing to remain weight stable throughout the study
* Free from alcohol dependence or abuse,
* Mini-mental stage examination score ≥21

Exclusion Criteria:

* Uncontrolled thyroid disease
* Regular vigorous aerobic (>6 bouts/week, >60 min/bout at a workload >6 METS)
* Blood donation within 8 weeks prior to enrolling in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in endothelial function at 3 months | 3 months
  Brachial artery flow-mediated dilation

SECONDARY OUTCOMES:
Change from baseline in suppression of endothelial function by mitochondrial oxidative stress at 3 months | 3 months
  Change in brachial artery flow-mediated dilation with acute, supratherapeutic MitoQ (160mg)
Change from baseline in aortic stiffness at 3 months | 3 months
  Carotid-femoral pulse wave velocity

OTHER OUTCOMES:
Change from baseline in serum exposure-induced endothelial cell reactive oxygen species production at 3 months | 3 months
  Endothelial cell whole-cell (CellROX) and mitochondria-specific (MitoSOX) reactive oxygen species levels after treatment with serum from subjects
Change from baseline in endothelial cell markers of oxidative stress and mitochondrial health from baseline at 3 months | 3 months
  Endothelial cell protein expression of nitrotyrosine and Fis1
Change from baseline in carotid artery stiffness at 3 months | 3 months
  Carotid artery beta-stiffness index
Change from baseline in circulating marker of oxidative stress at 3 months | 3 months
  Oxidized LDL levels in blood
Change from baseline in cerebrovascular reactivity at 3 months | 3 months
  Change in middle cerebral artery blood velocity in response to hypercapnia
Change from baseline in mitochondrial oxidative stress-mediated suppression of cerebrovascular reactivity at 3 months | 3 months
  Assessed as the change in cerebrovascular reactivity to hypercapnia following administration of a supratherapeutic dose of MitoQ known to scavenge mitochondrial reactive oxygen species
Change from baseline in internal carotid artery dilation at 3 months | 3 months
  Dilation of the internal carotid artery in response to hypercapnia
Change from baseline in mitochondrial oxidative stress-mediated suppression of internal carotid artery dilation at 3 months | 3 months
  Assessed as the change in internal carotid artery dilation to hypercapnia following administration of a supratherapeutic dose of MitoQ known to scavenge mitochondrial reactive oxygen species
Change from baseline in total cerebral blood flow at 3 months | 3 months
  Total cerebral blood flow
Change from baseline in serum exposure-induced brain endothelial cell nitric oxide and mitochondrial reactive oxygen species production at 3 months | 3 months
  Brain endothelial cell acetylcholine-induced nitric oxide production (DAR-4M-AM) and mitochondria-specific (MitoSOX) reactive oxygen species levels after treatment with serum from subjects

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Seals, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

REFERENCES:
- [Derived] Oh ES, Opoku G, Darvish S, Craighead DH, Ostrow A, Rossman MJ, Steele CN, Struemph T, You Z, Seals DR, Chonchol M, Nowak KL. Sex Differences in Dementia and Mild Cognitive Impairment in Nondialysis CKD. Clin J Am Soc Nephrol. 2025 Nov 20. doi: 10.2215/CJN.0000000922. Online ahead of print. No abstract available. PMID 41264372
- [Derived] Murray KO, Berryman-Maciel M, Darvish S, Coppock ME, You Z, Chonchol M, Seals DR, Rossman MJ. Mitochondrial-targeted antioxidant supplementation for improving age-related vascular dysfunction in humans: A study protocol. Front Physiol. 2022 Sep 15;13:980783. doi: 10.3389/fphys.2022.980783. eCollection 2022. PMID 36187760